CLINICAL TRIAL: NCT06577051
Title: Evaluation of Eustachian Tube Function With 226 and 1000 Hz Probes in Children Undergoing Tonsillectomy ± Adenoidectomy Without Tubal Dysfunction
Brief Title: Evaluation of Eustachian Tube Function With 226 and 1000 Hz Probes in Children Undergoing Tonsillectomy ± Adenoidectomy
Status: Completed | Type: Observational
Sponsor: Sumeyra DOLUOGLU (Other)
Responsible Party: Sponsor-Investigator, Sumeyra DOLUOGLU, M.D., Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Other Study IDs: SumeyraDoluoglu
Record Dates: First submitted 2024-08-21; First posted 2024-08-29 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Tonsillar Hypertrophy; Eustachian Tube Dysfunction; Tympanic Membrane Disorder; Eustachian Tube Dysfunction of Both Ears
Keywords: Eustachian tube; Tubal dysfunction; Tympanometry; High-frequency tympanometry; Eustachian tube dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children undergoing tonsillectomy ± adenoidectomy without tubal dysfunction: * 4-15 years old child patient
  * No preoperative tubal dysfunction detected in the patient
  * Willingness to participate in the study by the patient and his/her parents
  * The patient has no craniofacial anomaly, genetic disorder, cleft palate-lip anomaly
  * No bleeding disorder or disease
  Interventions: Diagnostic Test: Eustachian tube function test with 226 and 1000 Hz probes

INTERVENTIONS:
Diagnostic Test: Eustachian tube function test with 226 and 1000 Hz probes — In children undergoing tonsillectomy ± adenoidectomy without eustachian dysfunction, tympanometry with 226 Hz and 1000 Hz probes, ipsi and contralateral acoustic reflexes with 226 Hz probe, eustachian function test with 226 Hz probe (automatic Williams test) and play audiometry in young children and pure tone audiometry in older children are aimed to control tubal functions in preoperative period, postoperative day 1 and week 2.

SUMMARY:
In children undergoing tonsillectomy ± adenoidectomy without eustachian dysfunction, the objective is to control tubal functions with tympanometry utilising probes at 226 Hz and 1000 Hz, as well as measuring the ipsilateral and contralateral acoustic reflexes with a 226 Hz probe. An eustachian function test with a 226 Hz probe (automatic Williams test) and play audiometry are to be conducted on young children, while pure tone audiometry is to be conducted on older children, in the preoperative period, on the first day after surgery and in the second week after surgery. The primary objective is to ascertain whether the tubal functions, which are hypothesised to be impaired on the first day, return at the latest in the second week, with all tests evaluating the eustachian tube both directly and indirectly. The secondary objective is to determine whether this recovery occurs earlier with the 226 Hz probe or the 1000 Hz probe.

ELIGIBILITY:
Inclusion Criteria:

* 4-15 years old child patient
* No preoperative tubal dysfunction detected in the patient
* Willingness to participate in the study by the patient and his/her parents
* The patient has no craniofacial anomaly, genetic disorder, cleft palate-lip anomaly
* No bleeding disorder or disease

Exclusion Criteria:

* <3 years old, >15 years old paediatric patient
* Tubal dysfunction detected preoperatively
* Not wanting to participate in the study at any stage of the study
* The patient has craniofacial anomaly, genetic disorder, cleft palate-lip anomaly
* Having a bleeding disorder or disease

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 4-15 years who underwent tonsillectomy ± adenoidectomy for chronic tonsillitis or sleep breathing disorder without eustachian tube dysfunction were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation the functionality of the eustachian tube with odiometric tests | 14 days
  Evaluation the functionality of the eustachian tube, which was presumed to be compromised on the initial post-adenotonsillectomy day, and ascertainment whether it had recuperated by the second week. Tympanometry with 226 and 1000 Hz probes, eustachian function test with 226 Hz probe, ipsi and contralateral acoustic reflexes with 226 Hz probe and pure tone-play audiometry were performed in all patients one day before the operation. All tests were repeated on postoperative day 1 before the patient was discharged. All tests were repeated at the 2nd postoperative week.

SECONDARY OUTCOMES:
Evaluation the functionality of the eustachian tube with tympanometry the 226 Hz and 1000 Hz probes | 21 days
  It was investigated which of the 226 Hz and 1000 Hz probes used in these tests detected earlier recovery findings.

CONTACTS AND LOCATIONS:
Overall Officials: Sumeyra Doluoglu, MD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Doluoglu S, Gazeloglu AZ, Ulger N, Camalan BV, Dagli M. Evaluation of Eustachian tube function with dynamic and static tests in children undergoing adenotonsillectomy: A prospective clinical study. Int J Pediatr Otorhinolaryngol. 2025 Sep;196:112488. doi: 10.1016/j.ijporl.2025.112488. Epub 2025 Jul 14. PMID 40663994